CLINICAL TRIAL: NCT01018511
Title: A Randomized, Double-blind, Parallel Group, Placebo Controlled, Multi-center Study of Fixed Dose Combinations of Solifenacin Succinate (6 mg and 9 mg) With Tamsulosin Hydrochloride OCAS 0.4 mg and Tamsulosin Hydrochloride OCAS 0.4 mg Monotherapy, in Male Subjects With Lower Urinary Tract Symptoms (LUTS) Associated With Benign Prostatic Hyperplasia (BPH) With a Substantial Storage Component
Brief Title: Study of Solifenacin Succinate and Tamsulosin Hydrochloride OCAS in Males With Lower Urinary Tract Symptoms
Acronym: Neptune
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 905-CL-055; 2008-001211-37 (Other: EudraCT)
Record Dates: First submitted 2009-11-19; First posted 2009-11-23 (Estimated); Results first posted 2015-12-17 (Estimated); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Benign Prostatic Hyperplasia; Lower Urinary Tract Symptoms
Keywords: EC905; Solifenacin succinate; Tamsulosin hydrochloride OCAS; Treatment; Benign Prostatic Hyperplasia; Vesomni; Lower Urinary Tract Symptoms
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms | interventions — Solifenacin Succinate; Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Participants received 3 tablets once a day for 12 weeks. Placebo tamsulosin hydrochloride oral controlled absorption system (OCAS) 0.4 mg tablet; Placebo fixed dose combination (FDC) tamsulosin hydrochloride/solifenacin succinate 0.4 mg/6 mg tablet; Placebo FDC tamsulosin hydrochloride/solifenacin succinate 0.4 mg/9 mg tablet
  Interventions: Drug: Placebo tamsulosin hydrochloride OCAS 0.4 mg; Drug: Placebo FDC tamsulosin hydrochloride/solifenacin succinate 0.4 mg/6 mg; Drug: Placebo FDC tamsulosin hydrochloride/solifenacin succinate 0.4 mg/9 mg
- TOCAS 0.4 mg (Active Comparator): Participants received 3 tablets once a day for 12 weeks. Tamsulosin hydrochloride OCAS (TOCAS) 0.4 mg tablet; Placebo FDC tamsulosin hydrochloride/solifenacin succinate 0.4 mg/6 mg tablet; Placebo FDC tamsulosin hydrochloride/solifenacin succinate 0.4 mg/9 mg tablet
  Interventions: Drug: Placebo FDC tamsulosin hydrochloride/solifenacin succinate 0.4 mg/6 mg; Drug: Placebo FDC tamsulosin hydrochloride/solifenacin succinate 0.4 mg/9 mg; Drug: tamsulosin hydrochloride OCAS 0.4 mg
- FDC 0.4 mg/6 mg (Experimental): Participants received 3 tablets once a day for 12 weeks. Placebo TOCAS 0.4 mg tablet; FDC tamsulosin hydrochloride/solifenacin succinate 0.4 mg/6 mg tablet; Placebo FDC tamsulosin hydrochloride/solifenacin succinate 0.4 mg/9 mg tablet
  Interventions: Drug: Placebo tamsulosin hydrochloride OCAS 0.4 mg; Drug: Placebo FDC tamsulosin hydrochloride/solifenacin succinate 0.4 mg/9 mg; Drug: tamsulosin hydrochloride/solifenacin succinate fixed dose combination (0.4 mg/6 mg)
- FDC 0.4 mg/9 mg (Experimental): Participants received 3 tablets once a day for 12 weeks. Placebo TOCAS 0.4 mg tablet; Placebo FDC tamsulosin hydrochloride/solifenacin succinate 0.4 mg/6 mg tablet; FDC tamsulosin hydrochloride/solifenacin succinate 0.4 mg/9 mg tablet
  Interventions: Drug: Placebo tamsulosin hydrochloride OCAS 0.4 mg; Drug: Placebo FDC tamsulosin hydrochloride/solifenacin succinate 0.4 mg/6 mg; Drug: tamsulosin hydrochloride/solifenacin succinate fixed dose combination (0.4 mg/9 mg)

INTERVENTIONS:
Drug: Placebo tamsulosin hydrochloride OCAS 0.4 mg — tablet
  Arms: FDC 0.4 mg/6 mg; FDC 0.4 mg/9 mg; Placebo
Drug: Placebo FDC tamsulosin hydrochloride/solifenacin succinate 0.4 mg/6 mg — tablet
  Arms: FDC 0.4 mg/9 mg; Placebo; TOCAS 0.4 mg
Drug: Placebo FDC tamsulosin hydrochloride/solifenacin succinate 0.4 mg/9 mg — tablet
  Arms: FDC 0.4 mg/6 mg; Placebo; TOCAS 0.4 mg
Drug: tamsulosin hydrochloride OCAS 0.4 mg — tablet
  Other Names: Harnal ®; Omnic®; Flomax®; YM617
  Arms: TOCAS 0.4 mg
Drug: tamsulosin hydrochloride/solifenacin succinate fixed dose combination (0.4 mg/6 mg) — tablet
  Other Names: Vesomni; EC905
  Arms: FDC 0.4 mg/6 mg
Drug: tamsulosin hydrochloride/solifenacin succinate fixed dose combination (0.4 mg/9 mg) — tablet
  Other Names: EC905
  Arms: FDC 0.4 mg/9 mg

SUMMARY:
Clinical study to examine the efficacy, safety and tolerability of combination therapy of tamsulosin hydrochloride and solifenacin succinate compared to monotherapy of tamsulosin hydrochloride in the treatment of males with LUTS associated with BPH with a substantial storage component.

ELIGIBILITY:
Inclusion Criteria:

* Voiding and storage symptoms diagnosed as LUTS associated with BPH for ≥ 3 months
* A total International Prostate Symptom Score (IPSS) of ≥13
* A maximum urinary flow rate of ≥4.0 mL/s and ≤12.0 mL/s, with voided volume of ≥120 mL during free flow
* A micturition frequency of ≥8 and at least 2 episodes of urgency with Patient Perception of the Intensity of Urgency Scale grade 3 or 4 per day on average on the 3 day micturition diary (at randomization)

Exclusion Criteria:

* Any significant Post Void Residual volume (>150 mL)
* A prostate with estimated weight ≥75 ml as assessed by transvesical or transrectal ultrasound
* Evidence of a symptomatic urinary tract infection

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1334 (Actual)
Dates: Start 2010-01-11 (Actual); Primary Completion 2011-03-01 (Actual); Study Completion 2011-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Global Development
Locations (100):
- Austria (3):
  - Innsbruck
  - Salzburg
  - Vienna
- Minsk, Belarus
- Belgium (10):
  - Antwerp
  - Assebroek
  - Brussels
  - Edegem
  - Ghent
  - Kortrijk
  - Leuven
  - Liège
  - Sint-Truiden
  - Turnhout
- Czechia (8):
  - Hradec Králové
  - Ostrava
  - Pilsen
  - Prague
  - Roudnice nad Labem
  - Uherské Hradiště
  - Ústí nad Labem
  - Zdar
- France (12):
  - Aix-en-Provence
  - Angers
  - Bordeaux
  - Colmar
  - Dijon
  - Lyon
  - Montluçon
  - Orléans
  - Paris
  - Pierre-Bénite
  - Rennes
  - Tours
- Germany (13):
  - Bad Ems
  - Bautzen
  - Eisleben Lutherstadt
  - Frankfurt
  - Hagenow
  - Halle
  - Hamburg
  - Henningsdorf
  - Hettstedt
  - Koblenz
  - Leipzig
  - Neustadt in Sachsen
  - Uetersen
- Hungary (7):
  - Budapest
  - Körmend
  - Nyíregyháza
  - Sopron
  - Szekszárd
  - Szentes
  - Tatabánya
- Italy (9):
  - Avellino
  - Bari
  - Bergamo
  - Catania
  - Catanzaro
  - Florence
  - Palermo
  - Treviglio
  - Turin
- Netherlands (9):
  - Amsterdam
  - Apeldoorn
  - Doetinchem
  - Eindhoven
  - Etten-Leur
  - Maastricht
  - Sneek
  - Tilburg
  - Winterswijk
- Poland (6):
  - Bielsko-Biala
  - Bydgoszcz
  - Krakow
  - Puławy
  - Warsaw
  - Więcbork
- Russia (2):
  - Moscow
  - Saint Petersburg
- Slovakia (6):
  - Nitra
  - Piešťany
  - Prešov
  - Skalica
  - Trenčín
  - Žilina
- United Kingdom (14):
  - Birmingham
  - Bristol
  - Cardiff
  - Chorley
  - Glasgow
  - Liverpool
  - Manchester
  - Northwood
  - Nottingham
  - Plymouth
  - Reading
  - Sheffield
  - Taunton
  - Torquay

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Background] van Kerrebroeck P, Chapple C, Drogendijk T, Klaver M, Sokol R, Speakman M, Traudtner K, Drake MJ; NEPTUNE Study Group. Combination therapy with solifenacin and tamsulosin oral controlled absorption system in a single tablet for lower urinary tract symptoms in men: efficacy and safety results from the randomised controlled NEPTUNE trial. Eur Urol. 2013 Dec;64(6):1003-12. doi: 10.1016/j.eururo.2013.07.034. Epub 2013 Aug 3. PMID 23932438
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/hcp/study.aspx?ID=38

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Prior to randomization, participants entered a single-blind placebo run-in period for 2 weeks and completed a 3-day micturition diary. After the placebo run-in period, participants' eligibility criteria were re-confirmed and the participants were then randomized into the double-blind treatment period of the study.
Period: Overall Study
Arm/Group | Placebo | TOCAS 0.4 mg | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg
Started | 341 | 327 | 339 | 327
Randomized and Treated | 341 | 326 | 338 | 324
Completed | 315 | 295 | 299 | 294
Not Completed | 26 | 32 | 40 | 33
Not completed — Not fulfilling eligibility criteria | 6 | 7 | 7 | 3
Not completed — Adverse Event | 5 | 9 | 13 | 10
Not completed — Lack of Efficacy | 4 | 1 | 1 | 2
Not completed — Withdrawal by Subject | 6 | 5 | 11 | 9
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 5 | 8 | 7 | 9
Not completed — Miscellaneous | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAF): participants who received at least 1 dose of double-blind study drug and had any data reported after the first dose; For study-specific: Full Analysis Set (FAS): participants who received at least 1 dose of double-blind study drug and had either a total IPSS or TUS at baseline and at least 1 postbaseline total IPSS or TUS
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | TOCAS 0.4 mg | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg | Total
Number analyzed (Participants) | 341 | 326 | 337 | 324 | 1328
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (8.41) | 65.1 (7.98) | 65.3 (8.39) | 65.5 (7.71) | 65.4 (8.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 341 | 326 | 337 | 324 | 1328
Race/Ethnicity, Customized [Number; unit: participants]
  White | 337 | 325 | 334 | 321 | 1317
  Black | 0 | 1 | 1 | 2 | 4
  Asian | 3 | 0 | 1 | 0 | 4
  Other | 1 | 0 | 1 | 1 | 3
Total International Prostate Symptom Score (IPSS) [Mean (Standard Deviation); unit: units on a scale] — FAS population excluding 5 patients with invalid questionnaires. The number of participants was 318; 297; 311; 299 per treatment arm, respectively. The IPSS is a validated global questionnaire to assess the degree of "bother" from urinary symptoms, based on answers to 7 questions concerning urinary symptoms: -Incomplete emptying of the bladder -Intermittency -Weak stream -Hesitancy -Frequency -Urgency -Nocturia Each question is assigned points from 0 to 5 indicating increasing severity of the symptom. Total score can range from 0 to 35 (mildly symptomatic to severely symptomatic).
  units on a scale | 19.0 (4.48) | 18.7 (4.63) | 18.3 (4.31) | 18.6 (4.31) | 18.6 (4.44)
IPSS voiding score [Mean (Standard Deviation); unit: units on a scale] — FAS population excluding 5 patients with invalid questionnaires. The number of participants was 318; 297; 312; 299 per treatment arm, respectively. The IPSS is a validated global questionnaire to assess the degree of "bother" from urinary symptoms based on answers to 7 questions. Each question is assigned points from 0 to 5 indicating increasing severity of the particular symptom. The voiding score is the sum of the responses to 4 voiding questions (incomplete emptying of the bladder, intermittency, weak stream, hesitancy) and ranges from 0 to 20 (mildly symptomatic to severely symptomatic).
  units on a scale | 10.0 (3.53) | 9.8 (3.63) | 9.7 (3.61) | 9.7 (3.63) | 9.8 (3.60)
IPSS storage score [Mean (Standard Deviation); unit: units on a scale] — FAS population excluding 5 patients with invalid questionnaires. The number of participants was 318; 297; 311; 301 per treatment arm, respectively. The IPSS is a validated global questionnaire to assess the degree of "bother" from urinary symptoms based on answers to 7 questions. Each question is assigned points from 0 to 5 indicating increasing severity of the particular symptom. The storage symptom score is the sum of the responses to 3 storage questions (frequency, urgency and nocturia) and ranges from 0 to 15 (mildly symptomatic to severely symptomatic).
  units on a scale | 9.0 (2.42) | 8.9 (2.33) | 8.6 (2.39) | 8.8 (2.36) | 8.8 (2.38)
IPSS Quality of Life (QoL) score [Mean (Standard Deviation); unit: units on a scale] — FAS population excluding 5 patients with invalid questionnaires. The number of participants was 318; 297; 313; 301 per treatment arm, respectively. The QoL assessment was a single question asking the participant how he would feel about tolerating his current level of symptoms for the rest of his life. The answers ranged from 0 to 6 (delighted to terrible).
  units on a scale | 4.1 (1.12) | 4.1 (1.07) | 4.0 (1.15) | 4.1 (1.08) | 4.1 (1.11)
Total Urgency Frequency Score (TUFS) (previously known as Total Urgency Score ([TUS]) [Mean (Standard Deviation); unit: units on a scale] — FAS population.The number of participants was 318; 299; 314; 302 per arm, respectively.The Patient Perception of the Intensity of Urgency Scale (PPIUS) is a validated scale completed as part of the micturition diary. For each micturition and/or incontinence episode, the participant rated the degree of associated urgency according to the following 5-point categorical scale: 0.No urgency; 1.Mild urgency; 2.Moderate urgency; 3.Severe urgency; 4.Urgency incontinence. TUFS/TUS was the sum of the PPIUS gradings from the 3-day diary divided by the number of days on which urgency grading was recorded.
  units on a scale | 27.15 (8.80) | 27.85 (9.02) | 26.97 (8.66) | 26.39 (8.34) | 27.09 (8.71)
Micturitions/24 hours [Mean (Standard Deviation); unit: micturitions] — FAS population. The number of participants was 319; 299; 314; 302 per treatment arm, respectively. A micturition is any voluntary urination, excluding episodes of incontinence only. The mean number of micturitions per 24 hours was calculated from data recorded by the participant in the micturition diary for the 3 days preceding each clinic visit.
  micturitions | 11.37 (2.52) | 11.68 (2.86) | 11.48 (2.61) | 11.23 (2.56) | 11.44 (2.64)
Volume voided/micturition [Mean (Standard Deviation); unit: mL] — FAS population. The number of participants was 319; 299; 314; 302 per treatment arm, respectively. A micturition is any voluntary urination, excluding episodes of incontinence only. The mean volume voided per micturition was calculated from data recorded by the participant in the micturition diary for the 3 days preceding each clinic visit.
  mL | 160.49 (47.24) | 158.80 (47.21) | 160.74 (47.60) | 167.35 (50.32) | 161.82 (48.14)
Urgency episodes/24 hours [Mean (Standard Deviation); unit: urgency episodes] — FAS population. The number of participants was 319; 299; 314; 302 per treatment arm, respectively. An urgency episode is defined as an episode of strong desire to void accompanied by fear of leakage or pain. The mean number of urgency episodes with PPIUS grade 3 (Severe urgency) or 4 (Urgency incontinence) per 24 hours was calculated from data recorded by the participant in the micturition diary for the 3 days preceding each clinic visit.
  urgency episodes | 5.47 (3.26) | 5.51 (3.27) | 5.28 (3.22) | 5.18 (3.09) | 5.36 (3.21)
Incontinence episodes/24 hours [Mean (Standard Deviation); unit: incontinence episodes] — FAS population. The number of participants was 89; 66; 77; 86 per treatment arm, respectively. An incontinence episode is defined as an episode with any involuntary loss of urine. The mean number of incontinence episodes per 24 hours was calculated from data recorded by the participant in the micturition diary for the 3 days preceding each clinic visit.
  incontinence episodes | 1.79 (2.27) | 1.82 (1.73) | 1.70 (1.74) | 1.60 (2.23) | 1.73 (2.03)
Urgency incontinence episodes/24 hours [Mean (Standard Deviation); unit: urgency incontinence episodes] — FAS population. The number of participants was 86; 59; 69; 80 per treatment arm, respectively. An urgency incontinence episode is defined as an episode with any involuntary leakage of urine accompanied by or immediately preceded by urgency. The mean number of urgency incontinence episodes with PPIUS grade 3 (Severe urgency) or 4 (Urgency incontinence) per 24 hours was calculated from data recorded by the participant in the micturition diary for the 3 days preceding each clinic visit.
  urgency incontinence episodes | 1.62 (1.86) | 1.90 (1.75) | 1.71 (1.59) | 1.60 (2.24) | 1.70 (1.89)
Nocturia episodes/24 hours [Mean (Standard Deviation); unit: nocturia episodes] — FAS population. The number of participants was 306; 287; 302; 291 per treatment arm, respectively. A nocturia episode is defined as waking up at night to void (i.e., any voiding associated with sleep disturbance between the time the participant goes to bed with the intention to sleep until the time the patient gets up in the morning with the intention to stay awake). The mean number of nocturia episodes per 24 hours was calculated from data recorded by the participant in the micturition diary for the 3 days preceding each clinic visit.
  nocturia episodes | 2.41 (1.31) | 2.50 (1.31) | 2.37 (1.19) | 2.41 (1.26) | 2.42 (1.27)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to End of Treatment in Total International Prostate Symptom Score
Description: The International Prostate Symptom Score (IPSS) is a validated global questionnaire to assess the degree of urinary symptoms, based on answers to 7 questions concerning urinary symptoms: •Incomplete emptying of the bladder •Intermittency •Weak stream •Hesitancy •Frequency •Urgency •Nocturia Each question is assigned points from 0 to 5 indicating increasing severity of the symptom. Total score can range from 0 to 35 (mildly symptomatic to severely symptomatic).
Time Frame: Baseline and Week 12
Population: Full Analysis Set (FAS)-participants who received at least 1 dose of double-blind study drug and had either a total IPSS or TUS at baseline and at least 1 postbaseline total IPSS or TUS. Excluded 5 participants with invalid questionnaires. Last Observation Carried Forward (LOCF) imputation was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | TOCAS 0.4 mg | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg
Number analyzed (Participants) | 316 | 297 | 312 | 297
units on a scale | -5.4 (0.41) | -6.2 (0.42) | -7.0 (0.41) | -6.5 (0.42)
Statistical Analysis 1: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/6 mg; The non-inferiority of FDC vs TOCAS on the change from baseline to end of treatment in total IPSS. A FDC was regarded successful if it showed superiority vs. placebo for total IPSS, noninferiority vs. TOCAS alone for total IPSS along with superiority vs. TOCAS alone for TUS; Test type: Non-Inferiority or Equivalence — Overall power was 90% power for non-inferiority vs placebo for total IPSS. Only the FDC(s) that succeeded in stage 1 were evaluated in stage 2 for total IPSS. If both FDCs succeeded in stage 1, then both FDCs proceeded to stage 2 and the Hochberg procedure was implemented at one-sided alpha = 0.025. If one FDC succeeded in stage 1, then only this FDC proceeded to stage 2 and the FDC vs. TOCAS alone for non-inferiority was assessed at one-sided alpha = 0.025/2 = 0.0125; p = 0.001, Mixed Models Analysis — The primary analysis was adjusted for multiplicity for IPSS using the Hochberg procedure involving 2 stages: Stage 1, superiority to placebo and Stage 2: non-inferiority to tamsulosin alone, with a switch to superiority where applicable; A mixed model, including treatment group and country as fixed factors, center as a random effect, and baseline as a covariate; Least Squares Mean Difference = -0.8, 97.5% CI 2-sided [-1.73 to 0.11], Standard Error of Mean 0.41
Statistical Analysis 2: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/9 mg; The non-inferiority of FDC vs. TOCAS on the change from baseline to end of treatment in total IPSS. A FDC was regarded successful if it showed superiority vs. placebo for total IPSS, noninferiority vs. TOCAS alone for total IPSS along with superiority vs. TOCAS alone for TUS; Test type: Non-Inferiority or Equivalence — Only the FDC(s) that succeeded in stage 1 were evaluated in stage 2 for total IPSS. If both FDCs succeeded in stage 1, then both FDCs proceeded to stage 2 and the Hochberg procedure was implemented at one-sided alpha = 0.025. If one FDC succeeded in stage 1, then only this FDC proceeded to stage 2 and the FDC vs. TOCAS alone for non-inferiority was assessed at one-sided alpha = 0.025/2 = 0.0125; p = 0.028, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = -0.3, 97.5% CI 2-sided [-1.22 to 0.64], Standard Error of Mean 0.41
Statistical Analysis 3: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/6 mg; The superiority of FDC vs. TOCAS on the change from baseline to end of treatment in total IPSS; Test type: Superiority or Other; p = 0.048, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/9 mg; The superiority of FDC vs. TOCAS on the change from baseline to end of treatment in total IPSS; Test type: Superiority or Other; p = 0.483, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs FDC 0.4 mg/6 mg; The superiority of the FDC vs placebo on the change from baseline to end of treatment in total IPSS. A FDC was regarded successful if it showed superiority vs. placebo for total IPSS, noninferiority vs. TOCAS alone for total IPSS along with superiority vs. TOCAS alone for TUS; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = -1.6, 95% CI 2-sided [-2.4 to -0.9], Standard Error of Mean 0.40
Statistical Analysis 6: Comparison: Placebo vs FDC 0.4 mg/9 mg; The superiority of the FDC vs. placebo on the change from baseline to end of treatment in total IPSS. A FDC was regarded successful if it showed superiority vs. placebo for total IPSS, noninferiority vs. TOCAS alone for total IPSS along with superiority vs. TOCAS alone for TUS; Test type: Superiority or Other; p = 0.006, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = -1.1, 95% CI 2-sided [-1.9 to -0.3], Standard Error of Mean 0.41
Statistical Analysis 7: Comparison: Placebo vs TOCAS 0.4 mg; The superiority of TOCAS vs. placebo on the change from baseline to end of treatment in total IPSS. With a sample size of 274 participants per arm, the overall power to meet this outcome measure was 97% power for superiority vs placebo for total IPSS; Test type: Superiority or Other; p = 0.039, Mixed Models Analysis — No adjustments for multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = -0.8, 95% CI 2-sided [-1.6 to -0.0], Standard Error of Mean 0.41

2. Primary Outcome: Change From Baseline to End of Treatment in Total Urgency Frequency Score (TUFS, Previously Known as Total Urgency Score [TUS])
Description: The Patient Perception of the Intensity of Urgency Scale (PPIUS) is a validated scale completed as part of the micturition diary. For each micturition and/or incontinence episode, the participant rated the degree of associated urgency according to the following 5-point categorical scale: - 0. No urgency; - 1. Mild urgency; - 2. Moderate urgency; - 3. Severe urgency; - 4. Urgency incontinence TUFS was calculated as the sum of the PPIUS gradings from the 3-day diary divided by the number of days on which urgency grading was recorded. Higher scores indicate more severe urgency.
Time Frame: Baseline and Week 12
Population: FAS population. LOCF imputation was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | TOCAS 0.4 mg | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg
Number analyzed (Participants) | 315 | 295 | 313 | 302
units on a scale | -4.4 (0.68) | -6.7 (0.69) | -8.1 (0.67) | -7.6 (0.69)
Statistical Analysis 1: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/6 mg; The superiority of FDC 0.4 mg/6 mg vs. TOCAS in the change from baseline to end of treatment in TUS. A FDC was regarded successful if it showed superiority vs. placebo for total IPSS, noninferiority vs. TOCAS alone for total IPSS along with superiority vs. TOCAS alone for TUS; Test type: Superiority or Other; p = 0.025, Mixed Models Analysis — The primary analysis was adjusted for multiplicity for TUS using the Hochberg procedure; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -1.4, 97.5% CI 2-sided [-2.9 to 0.0], Standard Error of Mean 0.64
Statistical Analysis 2: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/9 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.162, Mixed Models Analysis — The primary analysis was adjusted for multiplicity for TUS using the Hochberg procedure; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -0.9, 97.5% CI 2-sided [-2.3 to 0.5], Standard Error of Mean 0.64
Statistical Analysis 3: Comparison: Placebo vs FDC 0.4 mg/6 mg; The superiority of FDC 0.4 mg/6 mg vs. placebo on the change from baseline to end of treatment in TUS; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = -3.7, 95% CI 2-sided [-4.9 to -2.5], Standard Error of Mean 0.62
Statistical Analysis 4: Comparison: Placebo vs FDC 0.4 mg/9 mg; The superiority of FDC 0.4 mg/9 mg vs. placebo on the change from baseline to end of treatment in TUS; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -3.2, 95% CI 2-sided [-4.4 to -1.9], Standard Error of Mean 0.63
Statistical Analysis 5: Comparison: Placebo vs TOCAS 0.4 mg; The superiority of TOCAS vs. placebo on the change from baseline to end of treatment in TUS; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -2.3, 95% CI 2-sided [-3.5 to -1.0], Standard Error of Mean 0.64

3. Secondary Outcome: Change From Baseline to End of Treatment in Mean Number of Micturitions Per 24 Hours
Description: A micturition is any voluntary urination, excluding episodes of incontinence only.The mean number of micturitions per 24 hours was calculated from data recorded by the participant in the micturition diary for the 3 days preceding each clinic visit.
Time Frame: Baseline and Week 12
Population: FAS population with data available at both baseline and end of treatment. LOCF imputation was used.
Measure: Least Squares Mean (Standard Error); unit: micturitions
Arm/Group | Placebo | TOCAS 0.4 mg | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg
Number analyzed (Participants) | 317 | 295 | 313 | 302
micturitions | -1.1 (0.16) | -1.7 (0.16) | -2.3 (0.16) | -1.9 (0.16)
Statistical Analysis 1: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/6 mg; Mean change vs TOCAS; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -0.6, 95% CI 2-sided [-1.0 to -0.3], Standard Error of Mean 0.17
Statistical Analysis 2: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/9 mg; Mean change vs TOCAS; Test type: Superiority or Other; p = 0.223, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -0.2, 95% CI 2-sided [-0.6 to 0.1], Standard Error of Mean 0.17
Statistical Analysis 3: Comparison: Placebo vs FDC 0.4 mg/6 mg; Mean change vs placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -1.2, 95% CI 2-sided [-1.5 to -0.8], Standard Error of Mean 0.17
Statistical Analysis 4: Comparison: Placebo vs FDC 0.4 mg/9 mg; Mean change vs placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -0.7, 95% CI 2-sided [-1.1 to -0.4], Standard Error of Mean 0.17
Statistical Analysis 5: Comparison: Placebo vs TOCAS 0.4 mg; Mean change vs placebo; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; least squares mean difference = -0.5, 95% CI 2-sided [-0.9 to -0.2], Standard Error of Mean 0.17

4. Secondary Outcome: Change From Baseline to End of Treatment in Mean Voided Volume Per Micturition
Description: A micturition is any voluntary urination, excluding episodes of incontinence only. The mean volume voided per micturition was calculated from data recorded by the participant in the micturition diary for the 3 days preceding each clinic visit.
Time Frame: Baseline and Week 12
Population: FAS population with data available at both baseline and end of treatment. LOCF imputation was used.
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Placebo | TOCAS 0.4 mg | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg
Number analyzed (Participants) | 317 | 295 | 313 | 302
mL | 11.1 (2.94) | 15.5 (3.02) | 38.6 (2.94) | 38.7 (3.01)
Statistical Analysis 1: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/6 mg; Mean change vs TOCAS; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 23.1, 95% CI 2-sided [16.6 to 29.6], Standard Error of Mean 3.33
Statistical Analysis 2: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/9 mg; Mean change vs TOCAS; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 23.2, 95% CI 2-sided [16.6 to 29.8], Standard Error of Mean 3.36
Statistical Analysis 3: Comparison: Placebo vs FDC 0.4 mg/6 mg; Mean change vs placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 27.4, 95% CI 2-sided [21.0 to 33.9], Standard Error of Mean 3.27
Statistical Analysis 4: Comparison: Placebo vs FDC 0.4 mg/9 mg; Mean change vs placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 27.6, 95% CI 2-sided [21.1 to 34.1], Standard Error of Mean 3.30
Statistical Analysis 5: Comparison: Placebo vs TOCAS 0.4 mg; Mean change vs placebo; Test type: Superiority or Other; p = 0.189, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 4.4, 95% CI 2-sided [-2.2 to 10.9], Standard Error of Mean 3.32

5. Secondary Outcome: Change From Baseline to End of Treatment in Maximum Volume Voided Per Micturition
Description: A micturition is any voluntary urination, excluding episodes of incontinence only. The maximum volume voided per micturition was calculated from data recorded by the participant in the micturition diary for the 3 days preceding each clinic visit.
Time Frame: Baseline and Week 12
Population: FAS population with data available at both baseline and end of treatment. LOCF imputation was used.
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Placebo | TOCAS 0.4 mg | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg
Number analyzed (Participants) | 317 | 295 | 313 | 302
mL | -5.9 (6.43) | -1.8 (6.62) | 12.7 (6.45) | 12.9 (6.63)
Statistical Analysis 1: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/6 mg; Mean change vs TOCAS; Test type: Superiority or Other; p = 0.053, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 14.5, 95% CI 2-sided [-0.2 to 29.3], Standard Error of Mean 7.51
Statistical Analysis 2: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/9 mg; Mean change vs TOCAS; Test type: Superiority or Other; p = 0.053, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 14.7, 95% CI 2-sided [-0.2 to 29.6], Standard Error of Mean 7.59
Statistical Analysis 3: Comparison: Placebo vs FDC 0.4 mg/6 mg; Mean change vs placebo; Test type: Superiority or Other; p = 0.012, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 18.5, 95% CI 2-sided [4.1 to 33.0], Standard Error of Mean 7.37
Statistical Analysis 4: Comparison: Placebo vs FDC 0.4 mg/9 mg; Mean change vs placebo; Test type: Superiority or Other; p = 0.012, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 18.7, 95% CI 2-sided [4.1 to 33.4], Standard Error of Mean 7.45
Statistical Analysis 5: Comparison: Placebo vs TOCAS 0.4 mg; Mean change vs placebo; Test type: Superiority or Other; p = 0.591, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 4.0, 95% CI 2-sided [-10.7 to 18.7], Standard Error of Mean 7.49

6. Secondary Outcome: Change From Baseline to End of Treatment in Mean Number of Urgency Episodes (PPIUS Grade 3 or 4) Per 24 Hours
Description: An urgency episode is defined as an episode of strong desire to void accompanied by fear of leakage or pain. The mean number of urgency episodes with PPIUS grade 3 (Severe urgency) or 4 (Urgency incontinence) per 24 hours was calculated from data recorded by the participant in the micturition diary for the 3 days preceding each clinic visit.
Time Frame: Baseline and Week 12
Population: FAS population and at least 1 urgency episode at baseline. LOCF imputation was used.
Measure: Least Squares Mean (Standard Error); unit: urgency episodes
Groups:
- FDC 0.4 mg 9 mg: Participants received 3 tablets once a day for 12 weeks. Placebo TOCAS 0.4 mg tablet; Placebo FDC tamsulosin hydrochloride/solifenacin succinate 0.4 mg/6 mg tablet; FDC tamsulosin hydrochloride/solifenacin succinate 0.4 mg/9 mg tablet
Arm/Group | Placebo | TOCAS 0.4 mg | FDC 0.4 mg/6 mg | FDC 0.4 mg 9 mg
Number analyzed (Participants) | 317 | 295 | 311 | 302
urgency episodes | -1.6 (0.24) | -2.5 (0.25) | -2.6 (0.24) | -2.8 (0.25)
Statistical Analysis 1: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/6 mg; Mean change vs TOCAS; Test type: Superiority or Other; p = 0.616, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -0.1, 95% CI 2-sided [-0.6 to 0.4], Standard Error of Mean 0.25
Statistical Analysis 2: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg 9 mg; Mean change vs TOCAS; Test type: Superiority or Other; p = 0.319, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -0.3, 95% CI 2-sided [-0.7 to 0.2], Standard Error of Mean 0.25
Statistical Analysis 3: Comparison: Placebo vs FDC 0.4 mg/6 mg; Mean change vs placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -1.0, 95% CI 2-sided [-1.5 to -0.6], Standard Error of Mean 0.24
Statistical Analysis 4: Comparison: Placebo vs FDC 0.4 mg 9 mg; Mean change vs placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -1.2, 95% CI 2-sided [-1.7 to -0.7], Standard Error of Mean 0.25
Statistical Analysis 5: Comparison: Placebo vs TOCAS 0.4 mg; Mean change vs placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -0.9, 95% CI 2-sided [-1.4 to -0.4], Standard Error of Mean 0.25

7. Secondary Outcome: Change From Baseline to End of Treatment in Mean Number of Urgency Incontinence Episodes Per 24 Hours
Description: An urgency incontinence episode is defined as an episode with any involuntary leakage of urine accompanied by or immediately preceded by urgency. The mean number of urgency incontinence episodes with PPIUS grade 3 (Severe incontinence) or 4 (Urgency incontinence) per 24 hours was calculated from data recorded by the participant in the micturition diary for the 3 days preceding each clinic visit.
Time Frame: Baseline and Week 12
Population: FAS population and at least 1 urgency incontinence episode at baseline. LOCF imputation was used.
Measure: Least Squares Mean (Standard Error); unit: urgency incontinence episodes
Arm/Group | Placebo | TOCAS 0.4 mg | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg
Number analyzed (Participants) | 86 | 57 | 69 | 80
urgency incontinence episodes | -1.0 (0.15) | -1.4 (0.18) | -1.3 (0.16) | -1.1 (0.16)
Statistical Analysis 1: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/6 mg; Mean change vs TOCAS; Test type: Superiority or Other; p = 0.591, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 0.1, 95% CI 2-sided [-0.3 to 0.5], Standard Error of Mean 0.22
Statistical Analysis 2: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/9 mg; Mean change vs TOCAS; Test type: Superiority or Other; p = 0.102, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 0.3, 95% CI 2-sided [-0.1 to 0.8], Standard Error of Mean 0.21
Statistical Analysis 3: Comparison: Placebo vs FDC 0.4 mg/6 mg; Mean change vs placebo; Test type: Superiority or Other; p = 0.204, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -0.2, 95% CI 2-sided [-0.6 to 0.1], Standard Error of Mean 0.19
Statistical Analysis 4: Comparison: Placebo vs FDC 0.4 mg/9 mg; Mean change vs placebo; Test type: Superiority or Other; p = 0.936, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 0.0, 95% CI 2-sided [-0.4 to 0.4], Standard Error of Mean 0.19
Statistical Analysis 5: Comparison: Placebo vs TOCAS 0.4 mg; Mean change vs placebo; Test type: Superiority or Other; p = 0.081, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -0.4, 95% CI 2-sided [-0.8 to 0.0], Standard Error of Mean 0.21

8. Secondary Outcome: Change From Baseline to End of Treatment in Mean Number of Incontinence Episodes Per 24 Hours
Description: An incontinence episode is defined as an episode with any involuntary loss of urine. The mean number of incontinence episodes per 24 hours was calculated from data recorded by the participant in the micturition diary for the 3 days preceding each clinic visit.
Time Frame: Baseline and Week 12
Population: FAS population and at least 1 incontinence episode at baseline. LOCF imputation was used.
Measure: Least Squares Mean (Standard Error); unit: incontinence episodes
Arm/Group | Placebo | TOCAS 0.4 mg | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg
Number analyzed (Participants) | 89 | 66 | 77 | 86
incontinence episodes | 0.1 (0.19) | -0.2 (0.22) | 0.0 (0.20) | 0.1 (0.19)
Statistical Analysis 1: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/6 mg; Mean change vs TOCAS; Test type: Superiority or Other; p = 0.511, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 0.2, 95% CI 2-sided [-0.3 to 0.6], Standard Error of Mean 0.24
Statistical Analysis 2: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/9 mg; Mean change vs TOCAS; Test type: Superiority or Other; p = 0.182, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 0.3, 95% CI 2-sided [-0.2 to 0.8], Standard Error of Mean 0.24
Statistical Analysis 3: Comparison: Placebo vs FDC 0.4 mg/6 mg; Mean change vs placebo; Test type: Superiority or Other; p = 0.552, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -0.1, 95% CI 2-sided [-0.6 to 0.3], Standard Error of Mean 0.22
Statistical Analysis 4: Comparison: Placebo vs FDC 0.4 mg/9 mg; Mean change vs placebo; Test type: Superiority or Other; p = 0.891, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 0.0, 95% CI 2-sided [-0.4 to 0.5], Standard Error of Mean 0.22
Statistical Analysis 5: Comparison: Placebo vs TOCAS 0.4 mg; Mean change vs placebo; Test type: Superiority or Other; p = 0.215, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -0.3, 95% CI 2-sided [-0.8 to 0.2], Standard Error of Mean 0.23

9. Secondary Outcome: Change From Baseline to End of Treatment in Mean Number of Nocturia Episodes Per 24 Hours
Description: A nocturia episode is defined as waking up at night to void (i.e., any voiding associated with sleep disturbance between the time the participant goes to bed with the intention to sleep until the time the patient gets up in the morning with the intention to stay awake). The mean number of nocturia episodes per 24 hours was calculated from data recorded by the participant in the micturition diary for the 3 days preceding each clinic visit.
Time Frame: Baseline and Week 12
Population: FAS population and at least 1 nocturia episode at baseline. LOCF imputation was used.
Measure: Least Squares Mean (Standard Error); unit: nocturia episodes
Arm/Group | Placebo | TOCAS 0.4 mg | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg
Number analyzed (Participants) | 282 | 256 | 275 | 271
nocturia episodes | -0.3 (0.07) | -0.4 (0.08) | -0.5 (0.07) | -0.4 (0.07)
Statistical Analysis 1: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/6 mg; Mean change vs TOCAS; Test type: Superiority or Other; p = 0.383, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -0.1, 95% CI 2-sided [-0.2 to 0.1], Standard Error of Mean 0.08
Statistical Analysis 2: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/9 mg; Mean change vs TOCAS; Test type: Superiority or Other; p = 0.402, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 0.1, 95% CI 2-sided [-0.1 to 0.2], Standard Error of Mean 0.08
Statistical Analysis 3: Comparison: Placebo vs FDC 0.4 mg/6 mg; Mean change vs placebo; Test type: Superiority or Other; p = 0.021, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -0.2, 95% CI 2-sided [-0.3 to -0.0], Standard Error of Mean 0.08
Statistical Analysis 4: Comparison: Placebo vs FDC 0.4 mg/9 mg; Mean change vs placebo; Test type: Superiority or Other; p = 0.584, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 0.0, 95% CI 2-sided [-0.2 to 0.1], Standard Error of Mean 0.08
Statistical Analysis 5: Comparison: Placebo vs TOCAS 0.4 mg; Mean change vs placebo; Test type: Superiority or Other; p = 0.166, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -0.1, 95% CI 2-sided [-0.3 to 0.0], Standard Error of Mean 0.08

10. Secondary Outcome: Change From Baseline to End of Treatment in Mean Number of Pads Used Per 24 Hours
Description: The mean number of pads per 24 hours was calculated from data recorded by the participant in the micturition diary for the 3 days preceding each clinic visit.
Time Frame: Baseline and Week 12
Population: FAS population and at least 1 use of a pad at baseline. LOCF imputation was used.
Measure: Least Squares Mean (Standard Error); unit: pads
Arm/Group | Placebo | TOCAS 0.4 mg | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg
Number analyzed (Participants) | 29 | 23 | 30 | 29
pads | -0.7 (0.23) | -0.8 (0.27) | -1.2 (0.24) | -1.2 (0.24)
Statistical Analysis 1: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/6 mg; Mean change vs TOCAS; Test type: Superiority or Other; p = 0.187, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -0.4, 95% CI 2-sided [-1.0 to 0.2], Standard Error of Mean 0.30
Statistical Analysis 2: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/9 mg; Mean change vs TOCAS; Test type: Superiority or Other; p = 0.203, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -0.4, 95% CI 2-sided [-1.0 to 0.2], Standard Error of Mean 0.31
Statistical Analysis 3: Comparison: Placebo vs FDC 0.4 mg/6 mg; Mean change vs placebo; Test type: Superiority or Other; p = 0.090, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -0.5, 95% CI 2-sided [-1.1 to 0.1], Standard Error of Mean 0.29
Statistical Analysis 4: Comparison: Placebo vs FDC 0.4 mg/9 mg; Mean change vs placebo; Test type: Superiority or Other; p = 0.098, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -0.5, 95% CI 2-sided [-1.1 to 0.1], Standard Error of Mean 0.29
Statistical Analysis 5: Comparison: Placebo vs TOCAS 0.4 mg; Mean change vs placebo; Test type: Superiority or Other; p = 0.772, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -0.1, 95% CI 2-sided [-0.7 to 0.5], Standard Error of Mean 0.31

11. Secondary Outcome: Change From Baseline to End of Treatment in IPSS Voiding Score
Description: The IPSS is a validated global questionnaire to assess the degree of urinary symptoms based on answers to 7 questions. Each question is assigned points from 0 to 5 indicating increasing severity of the particular symptom. The voiding score is the sum of the responses to 4 voiding questions (incomplete emptying of the bladder, intermittency, weak stream, hesitancy) and ranges from 0 to 20 (mildly symptomatic to severely symptomatic).
Time Frame: Baseline and Week 12
Population: FAS population with the exclusion of 5 participants with invalid questionnaires. LOCF imputation was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | TOCAS 0.4 mg | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg
Number analyzed (Participants) | 316 | 297 | 312 | 297
units on a scale | -3.0 (0.27) | -3.3 (0.28) | -3.7 (0.27) | -3.2 (0.28)
Statistical Analysis 1: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/6 mg; Mean change vs TOCAS; Test type: Superiority or Other; p = 0.210, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -0.3, 95% CI 2-sided [-0.9 to 0.2], Standard Error of Mean 0.27
Statistical Analysis 2: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/9 mg; Mean change vs TOCAS; Test type: Superiority or Other; p = 0.775, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 0.1, 95% CI 2-sided [-0.5 to 0.6], Standard Error of Mean 0.28
Statistical Analysis 3: Comparison: Placebo vs FDC 0.4 mg/6 mg; Mean change vs placebo; Test type: Superiority or Other; p = 0.010, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -0.7, 95% CI 2-sided [-1.2 to -0.2], Standard Error of Mean 0.27
Statistical Analysis 4: Comparison: Placebo vs FDC 0.4 mg/9 mg; Mean change vs placebo; Test type: Superiority or Other; p = 0.317, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -0.3, 95% CI 2-sided [-0.8 to 0.3], Standard Error of Mean 0.27
Statistical Analysis 5: Comparison: Placebo vs TOCAS 0.4 mg; Mean change vs placebo; Test type: Superiority or Other; p = 0.196, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -0.4, 95% CI 2-sided [-0.9 to 0.2], Standard Error of Mean 0.27

12. Secondary Outcome: Change From Baseline to End of Treatment in IPSS Storage Score
Description: The IPSS is a validated global questionnaire to assess the degree of urinary symptoms based on answers to 7 questions concerning urinary symptoms. Each question is assigned points from 0 to 5 indicating increasing severity of the particular symptom. The storage symptom score is the sum of the responses to 3 storage questions (frequency, urgency and nocturia) and ranges from 0 to 15 (mildly symptomatic to severely symptomatic).
Time Frame: Baseline and Week 12
Population: FAS population with the exclusion of 5 participants with invalid questionnaires. LOCF imputation was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | TOCAS 0.4 mg | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg
Number analyzed (Participants) | 316 | 297 | 312 | 297
units on a scale | -2.4 (0.20) | -2.9 (0.20) | -3.5 (0.20) | -3.3 (0.21)
Statistical Analysis 1: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/6 mg; Mean change vs TOCAS; Test type: Superiority or Other; p = 0.009, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -0.5, 95% CI 2-sided [-0.9 to -0.1], Standard Error of Mean 0.20
Statistical Analysis 2: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/9 mg; Mean change vs TOCAS; Test type: Superiority or Other; p = 0.045, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -0.4, 95% CI 2-sided [-0.8 to -0.0], Standard Error of Mean 0.21
Statistical Analysis 3: Comparison: Placebo vs FDC 0.4 mg/6 mg; Mean change vs placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -1.1, 95% CI 2-sided [-1.4 to -0.7], Standard Error of Mean 0.20
Statistical Analysis 4: Comparison: Placebo vs TOCAS 0.4 mg; Mean change vs placebo; Test type: Superiority or Other; p = 0.011, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -0.5, 95% CI 2-sided [-0.9 to -0.1], Standard Error of Mean 0.20
Statistical Analysis 5: Comparison: Placebo vs FDC 0.4 mg/9 mg; Mean change vs placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares men difference = -0.9, 95% CI 2-sided [-1.3 to -0.5], Standard Error of Mean 0.20

13. Secondary Outcome: Change From Baseline to End of Treatment in IPSS QoL Score
Description: The QoL assessment was a single question asking the participant how he would feel about tolerating his current level of symptoms for the rest of his life. The answers ranged from 0 to 6 (delighted to terrible).
Time Frame: Baseline and Week 12
Population: FAS population with the exclusion of 5 participants with invalid questionnaires. LOCF imputation was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | TOCAS 0.4 mg | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg
Number analyzed (Participants) | 316 | 297 | 312 | 297
units on a scale | -0.9 (0.11) | -1.0 (0.11) | -1.3 (0.11) | -1.3 (0.11)
Statistical Analysis 1: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/6 mg; Mean change vs TOCAS; Test type: Superiority or Other; p = 0.008, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; least squares mean difference = -0.3, 95% CI 2-sided [-0.5 to -0.1], Standard Error of Mean 0.10
Statistical Analysis 2: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/9 mg; Mean change vs TOCAS; Test type: Superiority or Other; p = 0.021, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -0.2, 95% CI 2-sided [-0.4 to -0.0], Standard Error of Mean 0.10
Statistical Analysis 3: Comparison: Placebo vs FDC 0.4 mg/6 mg; Mean change vs placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -0.4, 95% CI 2-sided [-0.6 to -0.2], Standard Error of Mean 0.10
Statistical Analysis 4: Comparison: Placebo vs FDC 0.4 mg/9 mg; Mean change vs placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -0.4, 95% CI 2-sided [-0.6 to -0.2], Standard Error of Mean 0.10
Statistical Analysis 5: Comparison: Placebo vs TOCAS 0.4 mg; Mean change vs placebo; Test type: Superiority or Other; p = 0.139, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -0.1, 95% CI 2-sided [-0.3 to 0.0], Standard Error of Mean 0.10

14. Secondary Outcome: Change From Baseline to End of Treatment in Individual IPSS Scores
Description: The IPSS is a validated global questionnaire to assess the degree of urinary symptoms, based on answers to 7 questions concerning urinary symptoms: •Incomplete emptying of the bladder •Intermittency •Weak stream •Hesitancy •Frequency •Urgency •Nocturia Each question is assigned points from 0 to 5 indicating increasing severity of the symptom.
Time Frame: Baseline and Week 12
Population: FAS population with the exclusion of 5 participants with invalid questionnaires. LOCF imputation was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | TOCAS 0.4 mg | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg
Number analyzed (Participants) | 316 | 297 | 312 | 297
units on a scale
  Incomplete emptying of the bladder | -0.9 (1.54) | -0.9 (1.52) | -1.0 (1.63) | -1.0 (1.48)
  Frequency | -1.0 (1.36) | -1.2 (1.42) | -1.3 (1.49) | -1.4 (1.41)
  Intermittency | -0.9 (1.41) | -0.8 (1.35) | -1.0 (1.47) | -0.7 (1.34)
  Urgency | -1.2 (1.55) | -1.3 (1.61) | -1.4 (1.51) | -1.6 (1.50)
  Weak stream | -1.1 (1.54) | -1.3 (1.57) | -1.3 (1.51) | -1.3 (1.56)
  Hesitancy | -0.5 (1.37) | -0.7 (1.26) | -0.8 (1.34) | -0.7 (1.29)
  Nocturia | -0.5 (1.23) | -0.7 (1.08) | -0.8 (1.08) | -0.6 (1.15)

15. Secondary Outcome: Change From Baseline to End of Treatment in Symptom Bother Score
Description: The Overactive Bladder Questionnaire (OAB-q) is a self-reported questionnaire with items relating to Symptom Bother and health-related quality of life (HRQoL). The Symptom Bother portion consists of an 8-item scale scored from 1 to 6. The total symptom bother score was calculated from the 8 answers and then transformed to range from 0 to 100, with 100 indicating worst severity. A negative change from baseline indicates an improvement.
Time Frame: Baseline and Week 12
Population: FAS population with data available at both baseline and end of treatment and the exclusion of 5 participants with invalid questionnaires. LOCF imputation was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | TOCAS 0.4 mg | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg
Number analyzed (Participants) | 315 | 297 | 312 | 297
units on a scale | -11.8 (1.26) | -14.4 (1.28) | -16.5 (1.26) | -17.1 (1.28)
Statistical Analysis 1: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/6 mg; Mean change vs TOCAS; Test type: Superiority or Other; p = 0.068, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -2.1, 95% CI 2-sided [-4.3 to 0.2], Standard Error of Mean 1.14
Statistical Analysis 2: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/9 mg; Mean change vs TOCAS; Test type: Superiority or Other; p = 0.020, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -2.7, 95% CI 2-sided [-4.9 to -0.4], Standard Deviation 1.15
Statistical Analysis 3: Comparison: Placebo vs FDC 0.4 mg/6 mg; Mean change vs placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -4.7, 95% CI 2-sided [-6.9 to -2.5], Standard Error of Mean 1.12
Statistical Analysis 4: Comparison: Placebo vs FDC 0.4 mg/9 mg; Mean change vs placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -5.3, 95% CI 2-sided [-7.5 to -3.1], Standard Error of Mean 1.13
Statistical Analysis 5: Comparison: Placebo vs TOCAS 0.4 mg; Mean change vs placebo; Test type: Superiority or Other; p = 0.022, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -2.6, 95% CI 2-sided [-4.8 to 0.4], Standard Error of Mean 1.14

16. Secondary Outcome: Change From Baseline to End of Treatment in Health Related QoL (HRQoL) Subscale: Coping Score
Description: The Overactive Bladder Questionnaire (OAB-q) is a self-reported questionnaire with items relating to Symptom Bother and health-related quality of life (HRQoL). The HRQoL portion consists of an 25-item HRQoL subscale containing the following domains scored from 1 to 6: - coping - concern - sleep - social interaction Coping score can range from 8 to 48 (none of the time to all of the time) and transformed to a scale from 0 to 100, with higher scores indicating better quality of life. A positive change from baseline indicates an improvement.
Time Frame: Baseline and Week 12
Population: as for outcome 15
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | TOCAS 0.4 mg | FDC 0.4 mg/6 mg | FDC 0.4 mg 9 mg
Number analyzed (Participants) | 315 | 297 | 312 | 297
units on a scale | 8.8 (1.24) | 11.0 (1.26) | 13.9 (1.24) | 13.4 (1.26)
Statistical Analysis 1: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/6 mg; Mean change vs TOCAS; Test type: Superiority or Other; p = 0.011, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 3.0, 95% CI 2-sided [0.7 to 5.2], Standard Error of Mean 1.16
Statistical Analysis 2: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg 9 mg; Mean change vs TOCAS; Test type: Superiority or Other; p = 0.035, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 2.5, 95% CI 2-sided [0.2 to 4.8], Standard Error of Mean 1.17
Statistical Analysis 3: Comparison: Placebo vs FDC 0.4 mg/6 mg; Mean change vs placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 5.1, 95% CI 2-sided [2.8 to 7.3], Standard Error of Mean 1.14
Statistical Analysis 4: Comparison: Placebo vs FDC 0.4 mg 9 mg; Mean change vs placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 4.6, 95% CI 2-sided [2.3 to 6.8], Standard Error of Mean 1.15
Statistical Analysis 5: Comparison: Placebo vs TOCAS 0.4 mg; Mean change vs placebo; Test type: Superiority or Other; p = 0.068, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 2.1, 95% CI 2-sided [-0.2 to 4.4], Standard Error of Mean 1.16

17. Secondary Outcome: Change From Baseline to End of Treatment in HRQoL Subscale: Concern Score
Description: The Overactive Bladder Questionnaire (OAB-q) is a self-reported questionnaire with items relating to Symptom Bother and health-related quality of life (HRQoL). The HRQoL portion consists of an 25-item HRQoL subscale containing the following domains scored from 1 to 6: •coping •concern •sleep •social interaction Concern score can range from 8 to 48 (none of the time to all of the time) and transformed to a scale from 0 to 100, with higher scores indicating better quality of life. A positive change from baseline indicates an improvement.
Time Frame: Baseline and Week 12
Population: as for outcome 15
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | TOCAS 0.4 mg | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg
Number analyzed (Participants) | 315 | 297 | 312 | 297
units on a scale | 7.5 (1.19) | 9.3 (1.21) | 12.0 (1.19) | 11.5 (1.21)
Statistical Analysis 1: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/6 mg; Mean change vs TOCAS; Test type: Superiority or Other; p = 0.013, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 2.6, 95% CI 2-sided [0.5 to 4.7], Standard Error of Mean 1.07
Statistical Analysis 2: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/9 mg; Mean change vs TOCAS; Test type: Superiority or Other; p = 0.043, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 2.2, 95% CI 2-sided [0.1 to 4.3], Standard Error of Mean 1.08
Statistical Analysis 3: Comparison: Placebo vs FDC 0.4 mg/6 mg; Mean change vs placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 4.4, 95% CI 2-sided [2.4 to 6.5], Standard Error of Mean 1.05
Statistical Analysis 4: Comparison: Placebo vs FDC 0.4 mg/9 mg; Mean change vs placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 4.0, 95% CI 2-sided [1.9 to 6.1], Standard Error of Mean 1.06
Statistical Analysis 5: Comparison: Placebo vs TOCAS 0.4 mg; Mean change vs placebo; Test type: Superiority or Other; p = 0.092, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 1.8, 95% CI 2-sided [-0.3 to 3.9], Standard Error of Mean 1.06

18. Secondary Outcome: Change From Baseline to End of Treatment in HRQoL Subscale: Sleep Score
Description: The Overactive Bladder Questionnaire (OAB-q) is a self-reported questionnaire with items relating to Symptom Bother and health-related quality of life (HRQoL). The HRQoL portion consists of an 25-item HRQoL subscale containing the following domains scored from 1 to 6: •coping •concern •sleep •social interaction Sleep score can range from 8 to 48 (none of the time to all of the time) and transformed to a scale from 0 to 100, with higher scores indicating better quality of life. A positive change from baseline indicates an improvement.
Time Frame: Baseline and Week 12
Population: as for outcome 15
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | TOCAS 0.4 mg | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg
Number analyzed (Participants) | 315 | 297 | 312 | 297
units on a scale | 8.3 (1.31) | 8.8 (1.33) | 11.9 (1.31) | 10.0 (1.33)
Statistical Analysis 1: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/6 mg; Mean change vs TOCAS; Test type: Superiority or Other; p = 0.011, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 3.1, 95% CI 2-sided [0.7 to 5.5], Standard Error of Mean 1.21
Statistical Analysis 2: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/9 mg; Mean change vs TOCAS; Test type: Superiority or Other; p = 0.314, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 1.2, 95% CI 2-sided [-1.2 to 3.6], Standard Error of Mean 1.23
Statistical Analysis 3: Comparison: Placebo vs FDC 0.4 mg/6 mg; Mean change vs placebo; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 3.6, 95% CI 2-sided [1.2 to 5.9], Standard Error of Mean 1.19
Statistical Analysis 4: Comparison: Placebo vs FDC 0.4 mg/9 mg; Mean change vs placebo; Test type: Superiority or Other; p = 0.161, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 1.7, 95% CI 2-sided [-0.7 to 4.1], Standard Error of Mean 1.21
Statistical Analysis 5: Comparison: Placebo vs TOCAS 0.4 mg; Mean change vs placebo; Test type: Superiority or Other; p = 0.708, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 0.5, 95% CI 2-sided [-1.9 to 2.8], Standard Error of Mean 1.21

19. Secondary Outcome: Change From Baseline to End of Treatment in HRQoL Subscale: Social Score
Description: The Overactive Bladder Questionnaire (OAB-q) is a self-reported questionnaire with items relating to Symptom Bother and health-related quality of life (HRQoL). The HRQoL portion consists of an 25-item HRQoL subscale containing the following domains scored from 1 to 6: •coping •concern •sleep •social interaction Social score can range from 8 to 48 (none of the time to all of the time) and transformed to a scale from 0 to 100, with higher scores indicating better quality of life. A positive change from baseline indicates an improvement.
Time Frame: Baseline and Week 12
Population: as for outcome 15
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | TOCAS 0.4 mg | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg
Number analyzed (Participants) | 315 | 297 | 312 | 297
units on a scale | 3.8 (0.96) | 4.5 (0.97) | 6.2 (0.95) | 5.8 (0.97)
Statistical Analysis 1: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/6 mg; Mean change vs TOCAS; Test type: Superiority or Other; p = 0.043, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 1.7, 95% CI 2-sided [0.1 to 3.3], Standard Error of Mean 0.83
Statistical Analysis 2: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/9 mg; Mean change vs TOCAS; Test type: Superiority or Other; p = 0.120, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 1.3, 95% CI 2-sided [-0.3 to 3.0], Standard Error of Mean 0.84
Statistical Analysis 3: Comparison: Placebo vs FDC 0.4 mg/6 mg; Mean change vs placebo; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 2.4, 95% CI 2-sided [0.8 to 4.0], Standard Error of Mean 0.82
Statistical Analysis 4: Comparison: Placebo vs FDC 0.4 mg/9 mg; Mean change vs placebo; Test type: Superiority or Other; p = 0.014, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 2.0, 95% CI 2-sided [0.4 to 3.7], Standard Error of Mean 0.83
Statistical Analysis 5: Comparison: Placebo vs TOCAS 0.4 mg; Mean change vs placebo; Test type: Superiority or Other; p = 0.384, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 0.7, 95% CI 2-sided [-0.9 to 2.4], Standard Error of Mean 0.83

20. Secondary Outcome: Change From Baseline to End of Treatment in HRQoL Subscale: Total Score
Description: The Overactive Bladder Questionnaire (OAB-q) is a self-reported questionnaire with items relating to Symptom Bother and health-related quality of life (HRQoL). The HRQoL portion consists of an 25-item HRQoL subscale containing the following domains scored from 1 to 6: •coping •concern •sleep •social interaction Total score is calculated by adding the 4 HRQoL subscale scores and transforming to a scale from 0 to 100, with higher scores indicating better quality of life. A positive change from baseline indicates an improvement.
Time Frame: Baseline and Week 12
Population: as for outcome 15
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | TOCAS 0.4 mg | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg
Number analyzed (Participants) | 315 | 297 | 312 | 297
units on a scale | 7.4 (1.06) | 8.8 (1.08) | 11.4 (1.06) | 10.7 (1.08)
Statistical Analysis 1: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/6 mg; Mean change vs TOCAS; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 2.6, 95% CI 2-sided [0.8 to 4.4], Standard Error of Mean 0.92
Statistical Analysis 2: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/9 mg; Mean change vs TOCAS; Test type: Superiority or Other; p = 0.035, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 2.0, 95% CI 2-sided [0.1 to 3.8], Standard Error of Mean 0.93
Statistical Analysis 3: Comparison: Placebo vs FDC 0.4 mg/6 mg; Mean change vs placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 4.0, 95% CI 2-sided [2.2 to 5.8], Standard Error of Mean 0.91
Statistical Analysis 4: Comparison: Placebo vs FDC 0.4 mg/9 mg; Mean change vs placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 3.3, 95% CI 2-sided [1.5 to 5.1], Standard Error of Mean 0.92
Statistical Analysis 5: Comparison: Placebo vs TOCAS 0.4 mg; Mean change vs placebo; Test type: Superiority or Other; p = 0.142, Mixed Models Analysis — No adjustments to multiplicity were made; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 1.4, 95% CI 2-sided [-0.5 to 3.2], Standard Error of Mean 0.92

21. Secondary Outcome: Percentage of Participants Who Were OAB-q Responders at End of Treatment
Description: A OAB-q responder was defined as a participant with an improvement from baseline in HRQoL subscale total score ≥ 10.
Time Frame: Week 12 (end of treatment)
Population: as for outcome 15
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TOCAS 0.4 mg | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg
Number analyzed (Participants) | 314 | 294 | 310 | 297
percentage of participants | 40.8 | 42.9 | 45.5 | 47.5
Statistical Analysis 1: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/6 mg; Difference vs TOCAS (superiority test); Test type: Superiority or Other; p = 0.874, Chi-squared — No adjustments for multiplicity were made
Statistical Analysis 2: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/9 mg; Difference vs TOCAS (superiority test); Test type: Superiority or Other; p = 0.240, Chi-squared — No adjustments for multiplicity were made
Statistical Analysis 3: Comparison: Placebo vs FDC 0.4 mg/6 mg; Difference vs placebo (superiority test); Test type: Superiority or Other; p = 0.324, Chi-squared — No adjustments for multiplicity were made
Statistical Analysis 4: Comparison: Placebo vs FDC 0.4 mg/9 mg; Difference vs placebo (superiority test); Test type: Superiority or Other; p = 0.043, Chi-squared — No adjustments for multiplicity were made
Statistical Analysis 5: Comparison: Placebo vs TOCAS 0.4 mg; Difference vs placebo (superiority test); Test type: Superiority or Other; p = 0.407, Chi-squared — No adjustments for multiplicity were made

22. Secondary Outcome: Change From Baseline to End of Treatment in EQ-5D Mobility Score
Description: The European quality of life-5 dimensions (EQ-5D) is an international standardized non-disease specific instrument for describing and valuing health status. The EQ5D has 5 domains: - mobility - self-care - usual activity - pain/discomfort - anxiety/depression Each domain has 3 response levels (1= no problem, 2= some problems, 3 = confined to bed).
Time Frame: Baseline and Week 12
Population: as for outcome 15
Measure: Number; unit: participants
Arm/Group | Placebo | TOCAS 0.4 mg | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg
Number analyzed (Participants) | 318 | 298 | 313 | 301
participants
  No problem -> No problem | 240 | 230 | 255 | 233
  No problem -> Some problem | 16 | 13 | 10 | 13
  No problem -> Confined to bed | 0 | 1 | 0 | 0
  No problem -> No data | 3 | 1 | 1 | 3
  Some problem -> No problem | 19 | 21 | 12 | 19
  Some problem -> Some problem | 40 | 31 | 35 | 31
  Some problem -> Confined to bed | 0 | 0 | 0 | 0
  Some problem -> No data | 0 | 0 | 0 | 1
  Confined to bed -> No problem | 0 | 0 | 0 | 0
  Confined to bed -> Some problem | 0 | 0 | 0 | 0
  Confined to bed -> Confined to bed | 0 | 0 | 0 | 0
  Confined to bed -> No data | 0 | 0 | 0 | 0
  No data -> No problem | 0 | 1 | 0 | 1
  No data -> Some problem | 0 | 0 | 0 | 0
  No data -> Confined to bed | 0 | 0 | 0 | 0
  No data -> No data | 0 | 0 | 0 | 0

23. Secondary Outcome: Change From Baseline to End of Treatment in EQ-5D Self-care Score
Description: The European quality of life-5 dimensions (EQ-5D) is an international standardized non-disease specific instrument for describing and valuing health status. The EQ5D has 5 domains: - mobility - self-care - usual activity - pain/discomfort - anxiety/depression Each domain has 3 response levels (1= no problem, 2= some problems, 3 = unable to wash/dress).
Time Frame: Baseline and Week 12
Population: as for outcome 15
Measure: Number; unit: participants
Arm/Group | Placebo | TOCAS 0.4 mg | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg
Number analyzed (Participants) | 318 | 298 | 313 | 301
participants
  No problem -> No problem | 295 | 273 | 293 | 286
  No problem -> Some problem | 8 | 8 | 3 | 4
  No problem -> Unable to wash/ dress | 0 | 0 | 0 | 0
  No problem -> No Data | 3 | 1 | 1 | 4
  Some problem -> No problem | 8 | 6 | 8 | 3
  Some problem -> Some problem | 3 | 8 | 6 | 3
  Some problem -> Unable to wash/ dress | 0 | 0 | 0 | 0
  Some problem -> No data | 0 | 0 | 0 | 0
  Unable to wash/ dress -> No problem | 0 | 0 | 1 | 0
  Unable to wash/ dress -> Some problem | 0 | 0 | 0 | 0
  Unable to wash/ dress -> Unable to wash/ dress | 0 | 1 | 0 | 0
  Unable to wash/ dress -> No data | 0 | 0 | 0 | 0
  No data -> No problem | 1 | 1 | 1 | 1
  No data -> Some problem | 0 | 0 | 0 | 0
  No data -> Unable to wash/ dress | 0 | 0 | 0 | 0
  No data -> No data | 0 | 0 | 0 | 0

24. Secondary Outcome: Change From Baseline to End of Treatment in EQ-5D Usual Activities Score
Description: The European quality of life-5 dimensions (EQ-5D) is an international standardized non-disease specific instrument for describing and valuing health status. The EQ5D has 5 domains: - mobility - self-care - usual activity - pain/discomfort - anxiety/depression Each domain has 3 response levels (1= no problem, 2= some problems, 3 = unable to perform usual activities).
Time Frame: Baseline and Week 12
Population: as for outcome 15
Measure: Number; unit: participants
Arm/Group | Placebo | TOCAS 0.4 mg | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg
Number analyzed (Participants) | 318 | 298 | 313 | 301
participants
  No problem -> No problem | 254 | 228 | 248 | 235
  No problem -> Some problem | 18 | 13 | 14 | 18
  No problem -> Unable to perform usual activities | 0 | 1 | 0 | 0
  No problem -> No data | 3 | 1 | 1 | 3
  Some problem -> No problem | 21 | 22 | 26 | 27
  Some problem -> Some problem | 22 | 28 | 22 | 17
  Some problem -> Unable to perform usual activities | 0 | 0 | 0 | 0
  Some problem -> No data | 0 | 0 | 0 | 1
  Unable to perform usual activities -> No problem | 0 | 1 | 2 | 0
  Unable to perform usual activities -> Some problem | 0 | 1 | 0 | 0
  Unable to perform usual activities -> same status | 0 | 1 | 0 | 0
  Unable to perform usual activities -> No data | 0 | 0 | 0 | 0
  No data -> No problem | 0 | 2 | 0 | 0
  No data -> Some problem | 0 | 0 | 0 | 0
  No data -> Unable to perform usual activities | 0 | 0 | 0 | 0
  No data -> No data | 0 | 0 | 0 | 0

25. Secondary Outcome: Change From Baseline to End of Treatment in EQ-5D Pain/Discomfort Score
Description: The European quality of life-5 dimensions (EQ-5D) is an international standardized non-disease specific instrument for describing and valuing health status. The EQ5D has 5 domains: - mobility - self-care - usual activity - pain/discomfort - anxiety/depression Each domain has 3 response levels (1= no pain, 2= moderate pain, 3 = extreme pain).
Time Frame: Baseline and Week 12
Population: as for outcome 15
Measure: Number; unit: participants
Arm/Group | Placebo | TOCAS 0.4 mg | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg
Number analyzed (Participants) | 318 | 298 | 313 | 301
participants
  No pain -> No pain | 162 | 159 | 153 | 152
  No pain -> Moderate pain | 14 | 14 | 19 | 24
  No pain -> Extreme pain | 2 | 1 | 1 | 0
  No pain -> No data | 3 | 0 | 1 | 2
  Moderate pain-> No pain | 55 | 41 | 61 | 41
  Moderate pain-> Moderate pain | 73 | 72 | 72 | 70
  Moderate pain-> Extreme pain | 2 | 2 | 1 | 1
  Moderate pain-> No data | 0 | 2 | 0 | 2
  Extreme pain -> No pain | 0 | 1 | 1 | 3
  Extreme pain -> Moderate pain | 4 | 2 | 2 | 4
  Extreme pain -> Extreme pain | 1 | 2 | 2 | 2
  Extreme pain -> No data | 0 | 0 | 0 | 0
  No data -> No pain | 0 | 2 | 0 | 0
  No data -> Moderate pain | 2 | 0 | 0 | 0
  No data -> Extreme pain | 0 | 0 | 0 | 0
  No data -> No data | 0 | 0 | 0 | 0

26. Secondary Outcome: Change From Baseline to End of Treatment in EQ-5D Anxiety/Depression Score
Description: The European quality of life-5 dimensions (EQ-5D) is an international standardized non-disease specific instrument for describing and valuing health status. The EQ5D has 5 domains: - mobility - self-care - usual activity - pain/discomfort - anxiety/depression Each domain has 3 response levels (1= not anxious, 2= moderately anxious, 3 = extremely anxious).
Time Frame: Baseline and Week 12
Population: as for outcome 15
Measure: Number; unit: participants
Arm/Group | Placebo | TOCAS 0.4 mg | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg
Number analyzed (Participants) | 318 | 298 | 313 | 301
participants
  Not anxious -> Not anxious | 219 | 213 | 233 | 214
  Not anxious -> Moderately anxious | 16 | 11 | 16 | 18
  Not anxious -> Extremely anxious | 0 | 0 | 0 | 0
  Not anxious -> No data | 3 | 0 | 1 | 3
  Moderately anxious -> Not anxious | 34 | 25 | 27 | 25
  Moderately anxious -> Moderately anxious | 42 | 43 | 39 | 34
  Moderately anxious -> Extremely anxious | 1 | 2 | 1 | 1
  Moderately anxious -> No data | 0 | 1 | 0 | 1
  Extremely anxious -> Not anxious | 2 | 0 | 1 | 0
  Extremely anxious -> Moderately anxious | 0 | 0 | 1 | 3
  Extremely anxious -> Extremely anxious | 1 | 2 | 3 | 2
  Extremely anxious -> No data | 0 | 0 | 0 | 0
  No data -> Not anxious | 0 | 1 | 1 | 0
  No data -> Moderately anxious | 0 | 0 | 0 | 0
  No data -> Extremely anxious | 0 | 0 | 0 | 0
  No data -> No data | 0 | 0 | 0 | 0

27. Secondary Outcome: Change From Baseline to End of Treatment in EQ-5D Visual Analogue Scale (VAS) Score
Description: Visual Analogue Scale (VAS) is part of the EQ-5D questionnaire. The VAS is self-rated by the participant ranging from 0 to 100 (worst imaginable health state to best imaginable health state).
Time Frame: Baseline and Week 12
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | TOCAS 0.4 mg | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg
Number analyzed (Participants) | 315 | 297 | 311 | 297
units on a scale | 4.0 (14.48) | 3.7 (12.69) | 5.5 (13.58) | 6.2 (15.52)

28. Secondary Outcome: Patient Global Impression Scale at End of Treatment: Overall Bladder Symptoms
Description: The Patient Global Impression (PGI) is a global questionnaire completed by the participant to assess both the change in the participants overall condition and the change in bladder symptoms since the start of the study. The questionnaire consists of 2 questions with 7 response levels ranging from 1 to 7 (very much improved to very much worse).
Time Frame: Baseline and Week 12
Population: as for outcome 15
Measure: Number; unit: participants
Arm/Group | Placebo | TOCAS 0.4 mg | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg
Number analyzed (Participants) | 318 | 298 | 313 | 301
participants
  Very Much Improved | 7 | 14 | 20 | 23
  Much Improved | 75 | 85 | 95 | 105
  Minimally Improved | 113 | 99 | 124 | 105
  No Change | 86 | 68 | 46 | 38
  Minimally Worse | 12 | 13 | 2 | 9
  Much Worse | 5 | 3 | 0 | 1
  Very Much Worse | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/6 mg; Difference vs TOCAS; Test type: Superiority or Other; p < .001, Chi-squared — No adjustments for multiplicity were made
Statistical Analysis 2: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/9 mg; Difference vs TOCAS; Test type: Superiority or Other; p < .001, Chi-squared — No adjustments for multiplicity were made
Statistical Analysis 3: Comparison: Placebo vs FDC 0.4 mg/6 mg; Difference vs placebo; Test type: Superiority or Other; p < .001, Chi-squared — No adjustments for multiplicity were made
Statistical Analysis 4: Comparison: Placebo vs FDC 0.4 mg/9 mg; Difference vs placebo; Test type: Superiority or Other; p < .001, Chi-squared — No adjustments for multiplicity were made
Statistical Analysis 5: Comparison: Placebo vs TOCAS 0.4 mg; Difference vs placebo; Test type: Superiority or Other; p = 0.058, Chi-squared — No adjustments for multiplicity were made

29. Secondary Outcome: Patient Global Impression Scale at End of Treatment: General Health
Description: as for outcome 28
Time Frame: Baseline and Week 12
Population: as for outcome 15
Measure: Number; unit: participants
Arm/Group | Placebo | TOCAS 0.4 mg | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg
Number analyzed (Participants) | 318 | 298 | 313 | 301
participants
  Very Much Improved | 5 | 9 | 10 | 7
  Much Improved | 43 | 58 | 72 | 75
  Minimally Improved | 79 | 77 | 87 | 94
  No Change | 152 | 126 | 110 | 94
  Minimally Worse | 15 | 9 | 8 | 10
  Much Worse | 2 | 3 | 0 | 1
  • Very Much Worse | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/6 mg; Difference vs TOCAS; Test type: Superiority or Other; p = 0.053, Chi-squared — No adjustments for multiplicity were made
Statistical Analysis 2: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/9 mg; Difference vs TOCAS; Test type: Superiority or Other; p = 0.031, Chi-squared — No adjustments for multiplicity were made
Statistical Analysis 3: Comparison: Placebo vs FDC 0.4 mg/6 mg; Difference vs placebo; Test type: Superiority or Other; p < .001, Chi-squared — No adjustments for multiplicity were made
Statistical Analysis 4: Comparison: Placebo vs FDC 0.4 mg/9 mg; Difference vs placebo; Test type: Superiority or Other; p < .001, Chi-squared — No adjustments for multiplicity were made
Statistical Analysis 5: Comparison: Placebo vs TOCAS 0.4 mg; Difference vs placebo; Test type: Superiority or Other; p = 0.018, Chi-squared — No adjustments for multiplicity were made

30. Secondary Outcome: Clinician Global Impression Scale at End of Treatment: Overall Bladder Symptoms
Description: The Clinician Global Impression (CGI) is a questionnaire completed by the physician to assess change in the participants bladder symptoms since the start of the study. The questionnaire consists of 1 question with 7 response levels ranging from 1 to 7 (very much improved to very much worse).
Time Frame: Baseline and Week 12
Population: as for outcome 15
Measure: Number; unit: participants
Arm/Group | Placebo | TOCAS 0.4 mg | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg
Number analyzed (Participants) | 318 | 298 | 313 | 301
participants
  Very Much Improved | 9 | 15 | 22 | 20
  Much Improved | 95 | 106 | 117 | 124
  Minimally Improved | 111 | 98 | 97 | 92
  No Change | 72 | 54 | 48 | 37
  Minimally Worse | 9 | 5 | 2 | 3
  Much Worse | 1 | 1 | 1 | 4
  Very Much Worse | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/6 mg; Difference vs TOCAS; Test type: Superiority or Other; p = 0.110, Chi-squared — No adjustments for multiplicity were made
Statistical Analysis 2: Comparison: TOCAS 0.4 mg vs FDC 0.4 mg/9 mg; Difference vs TOCAS; Test type: Superiority or Other; p = 0.071, Chi-squared — No adjustments for multiplicity were made
Statistical Analysis 3: Comparison: Placebo vs FDC 0.4 mg/6 mg; Difference vs placebo; Test type: Superiority or Other; p < .001, Chi-squared — No adjustments for multiplicity were made
Statistical Analysis 4: Comparison: Placebo vs FDC 0.4 mg/9 mg; Difference vs placebo; Test type: Superiority or Other; p < .001, Chi-squared — No adjustments for multiplicity were made
Statistical Analysis 5: Comparison: Placebo vs TOCAS 0.4 mg; Difference vs placebo; Test type: Superiority or Other; p = 0.019, Chi-squared — No adjustments for multiplicity were made

31. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Safety is monitored by collecting AEs, which include abnormal laboratory parameters, vital signs or ECG data if the abnormality induced clinical signs or symptoms, needed active intervention, interruption or discontinuation of study medication or was clinically significant. A serious AE (SAE) was an event resulting in death, persistent or significant disability/incapacity or congenital anomaly or birth defect, was life-threatening, required or prolonged hospitalization or was considered medically important. AEs were assessed by the Investigator for intensity as mild (no disruption of normal daily activities), moderate (affected normal daily activities) or severe (inability to perform daily activities) and for causal relationship to study drug. A treatment-emergent adverse event (TEAE) was defined as an AE that occurred after administration of the first dose of double-blind study drug until 14 days after the last dose of double-blind study drug.
Time Frame: From first dose of double-blind study drug up to 14 days of last dose of double-blind study drug (up to 14 weeks)
Population: Safety Analysis Set (SAF) - consisted of participants who received at least one dose of double blind study drug and for whom any data was reported after intake of the first dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | TOCAS 0.4 mg | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg
Number analyzed (Participants) | 341 | 326 | 337 | 324
participants
  Total TEAEs | 87 | 74 | 99 | 100
  Mild TEAEs | 59 | 42 | 68 | 68
  Moderate TEAEs | 25 | 29 | 27 | 27
  Severe TEAEs | 3 | 3 | 4 | 5
  Drug-related TEAEs | 30 | 27 | 57 | 65
  SAEs | 3 | 10 | 5 | 9
  Deaths | 0 | 1 | 1 | 0
  AEs Leading to Discontin | 5 | 9 | 13 | 10
  Drug-related AEs Leading to Discontin | 3 | 5 | 9 | 8

32. Secondary Outcome: Change From Baseline to End of Treatment in Post Void Residual (PVR) Volume
Description: PVR volume is the volume of urine retained after voiding. PVR volume was assessed by ultrasonography or bladder scan.
Time Frame: Baseline and Week 12
Population: SAF population with at least one baseline and one post-baseline PVR volume measured.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Placebo | TOCAS 0.4 mg | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg
Number analyzed (Participants) | 332 | 321 | 329 | 316
mL | -6.1 (36.39) | -5.0 (38.22) | 3.8 (45.39) | 12.3 (46.61)

33. Secondary Outcome: Change From Baseline to End of Treatment in Maximum Flow Rate (Qmax)
Description: Qmax during a micturition (urination) was recorded using uroflowmetry.
Time Frame: Baseline and Week 12
Population: SAF population with at least one baseline and one post-baseline micturition episode.
Measure: Mean (Standard Deviation); unit: mL/s
Arm/Group | Placebo | TOCAS 0.4 mg | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg
Number analyzed (Participants) | 306 | 289 | 305 | 290
mL/s | 3.3 (4.69) | 3.2 (4.62) | 3.8 (5.30) | 3.5 (5.35)

34. Secondary Outcome: Change From Baseline to End of Treatment in Average Flow Rate (Qmean)
Description: Qmean during a micturition (urination) was recorded using uroflowmetry.
Time Frame: Baseline and Week 12
Population: SAF population with at least one baseline and one post-baseline micturition episode.
Measure: Mean (Standard Deviation); unit: mL/s
Arm/Group | Placebo | TOCAS 0.4 mg | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg
Number analyzed (Participants) | 306 | 288 | 305 | 290
mL/s | 1.5 (2.61) | 1.3 (2.16) | 1.9 (2.75) | 1.7 (2.98)

35. Secondary Outcome: Apparent Clearance (CL/F) of Tamsulosin
Time Frame: Week 4, Week 8 and Week 12
Population: Pharmacokinetics Analysis Set (PKAS)- randomized participants who received at least 1 dose of double-blind study drug and had at least 1 quantifiable plasma concentration of tamsulosin OCAS and/or solifenacin. "N" indicates the number of participants with available data at each timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | TOCAS 0.4 mg | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg
Number analyzed (Participants) | 305 | 319 | 307
L/h
  Week 4 [N=263; 281; 274] | 2.78 (84.8) | 2.61 (85.8) | 2.53 (79.3)
  Week 8 [N=255; 259; 248] | 2.62 (79.0) | 2.41 (79.5) | 2.36 (93.3)
  Week 12 [N=163; 167; 166] | 2.52 (85.3) | 2.40 (74.1) | 2.46 (85.9)

36. Secondary Outcome: Maximum Concentration at Steady State (Cmaxss) of Tamsulosin
Time Frame: Week 4, Week 8 and Week 12
Population: PKAS population. "N" indicates the number of participants with available data at each timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | TOCAS 0.4 mg | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg
Number analyzed (Participants) | 305 | 319 | 307
ng/mL
  Week 4 [N= 263; 281; 274] | 7.38 (82.8) | 7.80 (94.3) | 8.00 (83.3)
  Week 8 [N= 255; 259; 248] | 7.69 (71.2) | 8.32 (73.4) | 8.46 (84.9)
  Week 12 [N= 163; 167; 166] | 7.97 (68.6) | 8.38 (69.0) | 8.16 (82.7)

37. Secondary Outcome: Minimum Concentration at Steady State (Cminss) of Tamsulosin
Time Frame: Week 4, Week 8 and Week 12
Population: PKAS population. "N" indicates the number of participants with available data at each timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | TOCAS 0.4 mg | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg
Number analyzed (Participants) | 305 | 319 | 307
ng/mL
  Week 4 [N= 263; 281; 274] | 4.19 (127.0) | 4.55 (146.0) | 4.75 (124.0)
  Week 8 [N= 255; 259; 248] | 4.63 (103.0) | 5.08 (106.0) | 5.19 (122.0)
  Week 12 [N= 163; 167; 166] | 4.84 (97.7) | 5.05 (96.2) | 4.94 (119.0)

38. Secondary Outcome: Time of Maximum Concentration at Steady State (Tmaxss) of Tamsulosin
Time Frame: Week 4, Week 8 and Week 12
Population: PKAS population. "N" indicates the number of participants with available data at each timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | TOCAS 0.4 mg | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg
Number analyzed (Participants) | 305 | 319 | 307
h
  Week 4 [N= 263; 281; 274] | 5.04 (4.1) | 5.06 (4.0) | 5.08 (3.6)
  Week 8 [N= 255; 259; 248] | 5.09 (3.4) | 5.10 (3.3) | 5.11 (3.4)
  Week 12 [N= 163; 167; 166] | 5.10 (3.6) | 5.09 (3.6) | 5.09 (3.3)

39. Secondary Outcome: Area Under the Curve at Steady State (AUCss) of Tamsulosin
Time Frame: Week 4, Week 8 and Week 12 (collection time points: trough, 1-3 hours post dose, 4-5 hours post-dose and 7-10 hours post-dose)
Population: PKAS population. "N" indicates the number of participants with available data at each timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/mL
Arm/Group | TOCAS 0.4 mg | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg
Number analyzed (Participants) | 305 | 319 | 307
ng.h/mL
  Week 4 [N= 263; 281; 274] | 144 (96.7) | 153 (111.0) | 158 (96.5)
  Week 8 [N= 255; 259; 248] | 153 (81.6) | 166 (84.0) | 169 (96.9)
  Week 12 [N= 163; 167; 166] | 159 (78.1) | 167 (77.4) | 162 (94.8)

40. Secondary Outcome: CL/F of Solifenacin
Time Frame: Week 4, Week 8 and Week 12
Population: PKAS population. "N" indicates the number of participants with available data at each timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg
Number analyzed (Participants) | 319 | 307
L/h
  Week 4 [N= 281;273] | 6.88 (53.6) | 7.00 (70.7)
  Week 8 [N= 258; 248] | 6.72 (51.7) | 6.67 (61.3)
  Week 12 [N= 166; 167] | 6.94 (59.3) | 6.87 (74.1)

41. Secondary Outcome: Cmaxss of Solifenacin
Time Frame: Week 4, Week 8 and Week 12
Population: PKAS population. "N" indicates the number of participants with available data at each timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg
Number analyzed (Participants) | 319 | 307
ng/mL
  Week 4 [N= 281; 273] | 29.4 (44.8) | 43.4 (51.4)
  Week 8 [N= 258; 248] | 30.0 (48.0) | 45.3 (48.5)
  Week 12 [N= 166; 167] | 29.1 (49.6) | 44.1 (50.7)

42. Secondary Outcome: Cminss of Solifenacin
Time Frame: Week 4, Week 8 and Week 12
Population: PKAS population. "N" indicates the number of participants with available data at each timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg
Number analyzed (Participants) | 319 | 307
ng/mL
  Week 4 [N= 281; 273] | 24.5 (50.5) | 36.1 (57.8)
  Week 8 [N= 258; 248] | 25.2 (54.1) | 38.2 (54.3)
  Week 12 [N= 166; 167] | 24.4 (55.6) | 37.0 (56.8)

43. Secondary Outcome: Tmaxss of Solifenacin
Time Frame: Week 4, Week 8 and Week 12
Population: PKAS population. "N" indicates the number of participants with available data at each timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg
Number analyzed (Participants) | 319 | 307
h
  Week 4 [N= 281; 273] | 5.47 (1.41) | 5.47 (1.2)
  Week 8 [N= 258; 248] | 5.48 (0.9) | 5.48 (0.9)
  Week 12 [N= 166; 167] | 5.48 (0.9) | 5.48 (0.9)

44. Secondary Outcome: AUCss of Solifenacin
Time Frame: as for outcome 39
Population: PKAS population. "N" indicates the number of participants with available data at each timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/mL
Arm/Group | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg
Number analyzed (Participants) | 319 | 307
ng.h/mL
  Week 4 [N= 281; 273] | 657 (46.8) | 970 (53.7)
  Week 8 [N= 258; 248] | 673 (50.3) | 1020 (50.7)
  Week 12 [N= 166; 167] | 652 (51.8) | 988 (53.0)

ADVERSE EVENTS:
Time Frame: From the first dose of double-blind study drug until 14 days after the last dose of double-blind study drug, up to 14 weeks.
Description: SAF population
Arm/Group | Placebo | TOCAS 0.4 mg | FDC 0.4 mg/6 mg | FDC 0.4 mg/9 mg
Serious Adverse Events (participants affected / at risk) | 3/341 | 10/326 | 5/337 | 9/324
Other Adverse Events (participants affected / at risk) | 5/341 | 3/326 | 36/337 | 43/324
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=341) | TOCAS 0.4 mg (N=326) | FDC 0.4 mg/6 mg (N=337) | FDC 0.4 mg/9 mg (N=324)
Urinary retention (Renal and urinary disorders) | 1 | 1 | 1 | 3
Angina unstable (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 0 | 1
Sick sinus syndrome (Cardiac disorders) | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 0 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Bronchiectasis (Infections and infestations) | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0
Cataract operation (Surgical and medical procedures) | 1 | 0 | 0 | 0
Gallbladder operation (Surgical and medical procedures) | 0 | 1 | 0 | 0
Hip arthroplasty (Surgical and medical procedures) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Varicose vein (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=341) | TOCAS 0.4 mg (N=326) | FDC 0.4 mg/6 mg (N=337) | FDC 0.4 mg/9 mg (N=324)
Constipation (Gastrointestinal disorders) | 1 | 1 | 12 | 18
Dry mouth (Gastrointestinal disorders) | 4 | 2 | 29 | 34

LIMITATIONS AND CAVEATS:
Company makes no warranties or representations of any kind as to the posting, expressed or implied, including warranties of merchantability and fitness for a particular purpose, and shall not be liable for any damages.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript at least 3 months prior to publication for review and comment. Sponsor may delay the publication to seek patent protection.